CLINICAL TRIAL: NCT04801251
Title: The Relation Between the Presence of Abnormal Clinical Cardiac Findings and Echocardiographic Findings in Newborn Infants
Brief Title: Red Flags for Cardiac Examination for Early Detection of Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sarah Bakry Gaber Ahmed, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Neonatal cardiology
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The relation between the presence of abnormal clinical cardiac findings and the abnormal echocardiographic findings
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resident (Other): Full history.complete systemic and cardiac physical examination
  Interventions: Diagnostic Test: Echocardiographic examination
- Assistant Lecturer (Other): Echocardiographic examination
  Interventions: Diagnostic Test: Echocardiographic examination

INTERVENTIONS:
Diagnostic Test: Echocardiographic examination — Each patient included will undergo full cardiac physical examination and echocardiographic examination
  Other Names: Full physical and cardiac examination

SUMMARY:
The study done to identify the relation between the presence of abnormal clinical cardiac findings and the echocardiographic findings in newborn infants.

DETAILED DESCRIPTION:
A full history will be taken, complete general systemic and cardiac examination will be done. All patients with abnormal physical cardiac examination in the neonatal period (≤ 28 days of age) according to the inclusion criteria will have echocardiographic examination.

ELIGIBILITY:
Inclusion Criteria:

* • Abnormal heart rate (< 90/min or < 160 per min )

  * Comfortable tachypnea ( RR > 60/min without other manifestations of respiratory distress)
  * Abnormal heart sounds (muffled, accentuated, single )
  * Abnormal precordial activity
  * Murmur: ( ≥ grade 3 intenisty, holosystolic timing, maximum intensity at upper left sternal border or with upright positing, diastolic murmur, harsh or blowing quality )
  * Abnormal oxygen saturation <90% in any extremity Oxygen saturation gradient > 3% difference in extremities.
  * Blood pressure gradient >10 mmHg higher in arms >10 mmHg lower in legs
  * Abnormal femoral pulses
  * Weakened pulses
  * Absent pulses
  * Hepatomegaly
  * Family history of cardiac disease

Exclusion Criteria:

* Newborns with disorders affecting the heart as anemia, septicemia, respiratory disorders as respiratory distress syndrome, pneumonia, hypoplastic lung, renal impairment, hypertension, metabolic disease, syndromatic CHF

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-10-20 (Estimated); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
Red flags for cardiac examination | 1 year
  A complete general systemic and cardiac examination will be done. All patients with abnormal physical cardiac examination in the neonatal period (≤ 28 days of age) according to the inclusion criteria will have echocardiographic examination.
  Methods:
  1. Echocardiogram reports will be reviewed and cardiovascular abnormalities will be noted. The presence of patent ductus arteriosus (PDA) will be considered a normal finding if present at ≤ 7 days of age but not beyond. A patent foramen ovale will be considered normal. A small muscular ventricular septal defect (VSD), although common in neonates and, will be considered an abnormal finding.
  2. All patients will have pulse oximeter screening, newborns with pulse oximetry ≥ 95% in the right hand or foot and ≤ 3% difference between the right hand and either foot at any time of testing have a normal result, and require no further testing.
The importance of history in detecting congenital heart disease | 1 year
  A full history will be taken, family history of congenital heart disease, mother's age and consanguinity, gravidity and parity should also be included.
  A File will be prepared for each neonate, which consist of demographic details including cardiac physical examination findings, birth weight, fetal age, history of folic acid intake by the mother, family history of cardiac disease, pulse oximeter screening, and results will be recorded.
  Data will be collected in form of taking history by interviewing questionnaire and full clinical examination will be done particularly cardiac examination and all findings will be recorded in patient clinical checklist.
  X^2 will be used to compare frequencies among different categories. Student T test, ANOVA will be used to test differences between means. ALL statistical analysis will be performed by using the SPSS version 20. P value <0.05 will be considered statistically significant for all applied statistical tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Ali, Professor, Study Director — Assiut University; Amira Shalaby, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: Yes
A full history will be taken, complete general systemic and cardiac examination will be done. All patients with abnormal physical cardiac examination in the neonatal period (≤ 28 days of age) according to the inclusion criteria will have echocardiographic examination.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting one year after publication
Access Criteria: all collected IPD, all IPD that underlie results in a publication

REFERENCES:
- [Result] Chitra N, Vijayalakshmi IB. Fetal echocardiography for early detection of congenital heart diseases. J Echocardiogr. 2017 Mar;15(1):13-17. doi: 10.1007/s12574-016-0308-2. Epub 2016 Aug 16. PMID 27530200
- [Result] Hiremath G, Kamat D. When to call the cardiologist: treatment approaches to neonatal heart murmur. Pediatr Ann. 2013 Aug;42(8):329-33. doi: 10.3928/00904481-20130723-13. No abstract available. PMID 23910039
- [Result] Triedman JK, Newburger JW. Trends in Congenital Heart Disease: The Next Decade. Circulation. 2016 Jun 21;133(25):2716-33. doi: 10.1161/CIRCULATIONAHA.116.023544. No abstract available. PMID 27324366
- See also: [Pediatric cardiology and congenital heart disease: from fetus to adult] — https://pubmed.ncbi.nlm.nih.gov/22269840/
- Available data/document: Study Protocol: Sarah bakry — https://www.outlook.com/aun.edu.eg — All data or information will be uploaded on the website